CLINICAL TRIAL: NCT02237170
Title: A Systems Biology Approach to Immune Monitoring in Patients With Castration-resistant Prostate Cancer Receiving SiPuleucel-T
Brief Title: Immune Monitoring on Sipuleucel-T
Acronym: PROVENGE
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 11-1689
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer
Keywords: Sipuleucel-T; Castration Resistant Prostate Cancer; Provenge
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Castration Resistant Metastatic Prostate Cancer: Castration Resistant Metastatic Prostate Cancer with no history of prior systemic chemotherapy

SUMMARY:
The purpose of this protocol is perform comprehensive immune monitoring studies in patients with castration-resistant prostate cancer receiving Sipuleucel-T in an effort to better understand the mechanism of action of this treatment.

DETAILED DESCRIPTION:
The primary objectives of this study are to:

1. Establish the phenotype and frequency of circulating immune cell compartments in patients undergoing treatment with Sipuleucel-T.
2. Determine the induction and the quality of prostate antigen-specific T cell immunity in patients undergoing treatment with Sipuleucel-T.
3. Correlate whole-blood RNA transcript-based signatures with clinical outcomes in patients treated with Sipuleucel-T.
4. Evaluate the cytokine and chemokine milieu in the peripheral blood pre- and post-treatment with Sipuleucel-T.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Written informed consent obtained
* Patients with castration-resistant prostate cancer who are initiating Sipuleucel-T as standard therapy
* No prior systemic chemotherapy for metastatic prostate cancer
* Hemoglobin > 9 mg/dl

Exclusion Criteria:

* Patients unable to understand the research protocol and/or provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from those patients who receive their care at Mount Sinai Medical Center, or a participating site
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Regulatory T cells (Tregs) | baseline and 1 year
  Establish the phenotype and frequency of circulating immune cell compartments in patients undergoing treatment with Sipuleucel-T looking at the change in regulatory T cells at 1 year post treatment compared to at baseline

SECONDARY OUTCOMES:
Change in Antigen Presenting Cells | baseline and 1 year
  Establish the phenotype and frequency of circulating immune cell compartments in patients undergoing treatment with Sipuleucel-T looking at the change in antigen presenting cells: DCs and B cells at 1 year post treatment compared to at baseline
Change in Prostate Antigen-specific T Cell Immunity | baseline and one year
Whole-blood RNA transcript-based signatures | baseline
  whole-blood RNA transcript-based signatures correlate with overall survival
Whole-blood RNA transcript-based signatures | up to 1 year
  whole-blood RNA transcript-based signatures correlate with overall survival
Change in cytokine milieu | baseline and 1 year
Change in chemokine milieu | baseline and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical College, New York, New York